CLINICAL TRIAL: NCT05245864
Title: Use of Blood Flow Restriction + Progressive Resistance Functional Training to Improve Functional Outcomes After Anterior Cruciate Ligament Reconstruction
Brief Title: Blood Flow Restriction Training in ACL Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty recruiting subjects; funding not renewed.
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 261865
Record Dates: First submitted 2022-01-26; First posted 2022-02-18 (Actual); Results first posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2023-03

CONDITIONS: Anterior Cruciate Ligament Injuries
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- physical therapy with blood flow restriction (Experimental)
  Interventions: Other: blood flow restriction
- physical therapy without blood flow restriction (Other): Standard of care.
  Interventions: Other: physical therapy standard of care

INTERVENTIONS:
Other: blood flow restriction — Blood flow to the legs will be mostly restricted temporarily during physical therapy exercises for the initial several weeks of physical therapy.
  Arms: physical therapy with blood flow restriction
Other: physical therapy standard of care — the current standard of care after surgery for ACL repair.
  Arms: physical therapy without blood flow restriction

SUMMARY:
This will be a randomized pilot study to determine the effectiveness of Personalized Blood Flow Restriction (PBFR) technique in conjunction with prescribed physical therapy (PT) in a cohort of anterior cruciate ligament (ACL) reconstruction subjects

DETAILED DESCRIPTION:
This will be a randomized pilot study to determine the effectiveness of Personalized Blood Flow Restriction (PBFR) technique in conjunction with prescribed physical therapy (PT) in a cohort of anterior cruciate ligament (ACL) reconstruction subjects. Both groups of subjects will undergo unilateral ACL reconstruction at University of Arkansas for Medical Sciences (UAMS), followed by prescribed PT at the UAMS Orthopedic Clinic at Colonel Glenn.

Up to 25 subjects will be enrolled. Half are randomized to the BFR group with the other will perform PT without BFR.

Data collection will occur at four approximate occasions: pre-surgery, 8-weeks postop, 12-weeks postop, and 16-weeks postop.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, ages 18-34 years.
2. Scheduled to undergo elective ACL surgery at UAMS.
3. Capable of providing informed consent.
4. Willing to exercise with BFR.
5. COVID-19 negative or asymptomatic.

Exclusion Criteria:

1. Any surgical indication other than ACL repair.
2. Body mass index >40.
3. Pregnant female.
4. Neurological, musculoskeletal, or other disorder that would preclude them from completing the exercise training intervention and all performance tests.
5. Hypertension as evidenced by systolic BP >150 at rest OR diastolic BP >85 at rest.
6. Heart failure as evidenced by use of prescription diuretics.
7. History of atrial fibrillation.
8. Oxygen saturation <95% on room air at rest.
9. Any other medical condition that would interfere with testing or increase one's risk of complications during exercise.
10. Currently receiving androgen (e.g., testosterone) or anabolic (e.g., GH, IGF-I) therapy.
11. Compromised vascular circulation in the legs (e.g. peripheral vascular disease).
12. History of deep vein thrombosis.
13. Varicose veins in the legs.
14. Known Sickle cell disease or trait.
15. Unwilling to avoid using protein or amino-acid supplements during participation.
16. Unwilling to avoid using BFR during prescribed post-operative physical therapy.

Ages: 18 Years to 34 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2022-04-18 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arny A Ferrando, Ph.D., Principal Investigator — University of Arkansas
Locations (1):
- UAMS Center on Aging, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Physical Therapy With Blood Flow Restriction | Physical Therapy Without Blood Flow Restriction
Started | 1 | 1
Completed | 0 | 0
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Physical Therapy With Blood Flow Restriction | Physical Therapy Without Blood Flow Restriction | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 0 | 1 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Maximal Voluntary Contraction
Description: Max torque produced in newton meter per second during an isometric contraction
Time Frame: 16-weeks post-surgery
Population: Participant who did Physical therapy without blood flow restriction completed only enrollment and pre testing. Participant who completed physical therapy with blood flow restriction completed only enrollment, pre testing, and one post operative testing visit.
Arm/Group | Physical Therapy With Blood Flow Restriction | Physical Therapy Without Blood Flow Restriction
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: ACL Repair Range of Motion
Description: Measured at the knee, therefore, the degree to which the lower limb can move around knee joint in relation to the upper limb.
Time Frame: from enrollment to the end of treatment at 16 weeks
Population: No participant completed this measure.
Arm/Group | Physical Therapy With Blood Flow Restriction | Physical Therapy Without Blood Flow Restriction
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 20 weeks
Arm/Group | Physical Therapy With Blood Flow Restriction | Physical Therapy Without Blood Flow Restriction
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-03): https://cdn.clinicaltrials.gov/large-docs/64/NCT05245864/Prot_SAP_000.pdf